CLINICAL TRIAL: NCT06720948
Title: An Observational Multicenter Consecutive Case Study of Long-Term Safety and Effectiveness Outcomes of a Real-World Population
Brief Title: The ION Facet Screw System Ambispective Evaluation
Acronym: FixatION
Status: Active, not recruiting | Type: Observational
Sponsor: SurGenTec LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: TSN-2024-001; ION Facet RWE Study (Other: SurGenTec)
Record Dates: First submitted 2024-11-21; First posted 2024-12-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Intra-facet ION 3D Facet Screw System
Keywords: ION; fixation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cervical: Previously implanted bilaterally intra-facet with the SurGenTec ION 3D Facet Screw System at one or two contiguous levels of the cervical spine (C3-C7)
  Interventions: Device: ION 3D Facet Screw System
- Lumbar: Previously implanted bilaterally intra-facet with the SurGenTec ION 3D Facet Screw System at one or two contiguous levels of the lumbar spine (L3-S1)
  Interventions: Device: ION 3D Facet Screw System

INTERVENTIONS:
Device: ION 3D Facet Screw System — Observational study of subjects previously implanted with ION 3D Facet Screw System.

SUMMARY:
The purpose of this observational, multi-center, ambispective, serial case study is to collect real-world patient outcomes that characterize the long-term safety and effectiveness of the SurGenTec ION 3D® Facet Screw System in a cervical spine and a lumbar spine application.

DETAILED DESCRIPTION:
The statistical analysis of the data obtained from this study will be performed using a validated statistical software program such as SPSS®. All tests will be performed at the 0.05 significance level, unless otherwise specified. Analysis will be based upon the treated population defined as all subjects that underwent standard of care surgical intervention with the SurGenTec ION 3D Facet Screw System that agreed to participate in this data collection initiative.

Data collected in this study will be documented using summary tables and subject data listings. Continuous variables will be summarized using descriptive statistics, specifically the mean, median, standard deviation, minimum, and maximum, and a 95% confidence interval for the mean based on the t-distribution. Categorical variables will be summarized using frequencies, percentages, and 95% confidence intervals for the true proportions. Resultant of the observational study design, this evaluation is not powered to test a hypothesis. It is designed to yield supplemental long-term information in this real-world population.

The analysis will be stratified by lumbar and cervical patients. Additionally, each cohort will evaluate the following analysis populations:

Enrolled Population: This dataset will include all subjects who were screened and enrolled into the study.

Evaluable Population: This dataset will exclude subjects with ION 3D Facet Screw device improperly placed

To minimize the introduction of bias into this observational low risk evaluation, the following measures will be observed:

* Complete and accurate prespecified data shall be obtained,
* All cervical and all lumbar patients at a study site that were previously implanted with the ION 3D Facet Screw System will be reviewed for possible study inclusion (all-comers study design),
* All participants will be enrolled under the same study entrance criteria,
* All participants shall follow the same prospectively designed study protocol,
* Serious Adverse Event adjudication will be performed by independent blinded reviewer, and
* Radiographic measurements and CT assessments will be performed by blinded independent core lab.

In consideration of the retrospective nature of this investigation coupled with a possible 1-time prospective evaluation, data monitoring will not be performed. However, data edits and database checks will be built into the EDC system to minimize the potential for data entry errors. Further, TSN, as the entity responsible for overall study conduct/management, will review all data entered and ensure appropriate source documentation is available to support data extraction/collection.

ELIGIBILITY:
Inclusion Criteria:

* Previously implanted intra-facet with one ION® Facet Screw placed per joint bilaterally at one or more contiguous levels of the cervical spine (C3-C7), or one or more contiguous levels of the lumbar spine (L3-S1),
* Must have supplemental fixation at the target level(s),
* Skeletally mature (minimum age of 21 years but not greater than 80 years),
* Be willing and able to comply with the study protocol requirements, and
* Be willing to sign the study-specific Informed Consent Document.

Exclusion Criteria:

* Implanted with the ION Facet Screw System at a spinal level that includes the thoracic spine (T1-T12),
* Unilateral fixation with the ION Fact Screw System,
* Current tobacco use
* Body Mass Index of >40,
* Current active or suspected malignancy, or a cancer diagnosis that was ongoing during the patient's treatment and healing period,
* Significant metabolic bone disease (diagnosis of osteoporosis or osteomalacia),
* Currently taking medications that are known to potentially interfere with bone healing (e.g. chronic oral/systemic steroids),
* Pregnant or nursing female, or
* Incarcerated at the time of the required 12-month evaluation.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients that have previously undergone a cervical or lumbar facet fusion with the ION® Facet Screw System (IFSS)
  * Patients must be a minimum of one year postoperative
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Quantitative Fusion | 12 Months Post-Op
  Defined as <5 degrees of angulation and/or <3mm translation as measured on dynamic flexion and extension radiographs
Rate of Stability of operative level(s) | 12 Months Post-Op
  Substantial motion defined as >5 degrees angulation and/or >3mm translation as measured on dynamic flexion and extension radiographs.
Rate of Qualitative Fusion | 12 Months Post-Op
  Bridging bone present external to the ION 3D facet screw device as observed on CT scan.
Incidence of Serious Adverse Events | 12 Months Post-Op
  Freedom from ION 3D facet screw device-related serious adverse events as adjudicate by an independent reviewer.
Incidence of Secondary Surgical Events | 12 Months Post-Op
  Secondary surgical events at the operative level(s) from intraoperative through ≥12-month evaluation timepoint.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orthopaedics Northeast, Fort Wayne, Indiana
  - Neuroscience Specialists, Oklahoma City, Oklahoma